CLINICAL TRIAL: NCT01863407
Title: A Phase 3, Multicenter, Double-Blind, Placebo-Controlled, Parallel Study of Dexamethasone-Allantoin-Metronidazole (DAM) Solution in the Treatment of Post-Operative Ileus (POI) in Subjects Undergoing Abdominal Operation
Brief Title: Study of Dexamethasone-Allantoin-Metronidazole (DAM) Solution in the Treatment of Post-Operative Ileus (POI)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Bozhiyin T&S Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BZY 001
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Postoperative Ileus
Keywords: Ileus; Intestinal Obstruction; Intestinal Diseases; Gastrointestinal Diseases; Digestive System Diseases
MeSH Terms: conditions — Ileus; Intestinal Obstruction; Intestinal Diseases; Gastrointestinal Diseases; Digestive System Diseases | interventions — Solutions; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DAM Solution (Experimental): Preheated to a temperature level, mixed the DAM Solution 2ml and Normal Saline 250ml, poured into abdominal cavity and infiltrate the operative field before the abdominal closure
  Interventions: Drug: DAM
- Normal Saline (Placebo Comparator): Preheated the Normal Saline 250ml to a temperature level, poured into abdominal cavity and infiltrate the operative field before the abdominal closure
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: DAM — composed of dexamethasone, allantoin and metronidazole
  Other Names: Dexamethasone-Allantoin-Metronidazole (DAM) Solution
  Arms: DAM Solution
Drug: Normal Saline — Normal Saline 250ml
  Other Names: NS
  Arms: Normal Saline

SUMMARY:
This study is being conducted to determine whether Dexamethasone-Allantoin-Metronidazole (DAM) Solution can accelerate recovery of gastrointestinal function following abdominal operation when compared with a placebo.

DETAILED DESCRIPTION:
Postoperative ileus (POI) is temporary slowing down or stopping of bowel function and a slowing down of movement of contents of the intestines. This functional impairment persists for a variable duration following surgery, usually resolving within 1 day in the small intestine, 1 to 3 days in the stomach and 3 to 5 days in the colon. When POI persists for more than 5 days, it is generally considered severe, sometimes referred to as complicated or prolonged POI, and increases the risk for related morbidity. This is a randomized, controlled, double-blind study designed to evaluate the tolerability and efficacy of DAM solution for the treatment of POI in patients following abdominal operation. It will be conducted at multiple centers in China. A total of 480 patients will be enrolled in the study. Patient participation in the study will last for up to postoperative day 7 [POD 7] , with follow-up safety assessments to occur 7 days after the operation.The treatment outcome measures include: 1) GI2(Time to achieve recovery of both upper and lower GI function as measured by a composite endpoint of time to the first bowel movement and time to tolerate first solid food). 2) Time to ready for discharge. 3) Time to the first flatus.

ELIGIBILITY:
Inclusion Criteria:

* are either Male or Female at least 18 years of age;
* Had an American Society of Anesthesiologists (ASA) Physical Status Score of I-III;
* Were scheduled to undergo partial small or large BR with primary anastomosis (performed completely by laparotomy); biliary-enteric Roux-en-Y anastomosis surgery;
* BMI (kg/m^2) index≥15 and ≤30;
* Understood the procedures, agreed to participate in the study program, and voluntarily signed the informed consent form.

Exclusion Criteria:

* Had complete bowel obstruction;
* Were scheduled for a total colectomy;
* Were scheduled for a ileal pouch-anal anastomosis;
* Were scheduled for a colostomy, ileostomy;
* Had a history of gastrectomy, total colectomy, gastric bypass, short bowel syndrome, or multiple previous abdominal surgeries;
* Had clinically significant laboratory abnormalities on screening(such as: ALT, AST were more than 2 times the upper limit of normal value; Cr is greater than 1.2 times the upper normal limit, according to the center for the study of the normal value range);
* Applied the intravenous or epidural postoperative analgesia pump;
* Bowel preparation does not meet the requirements;
* Were allergy to components of the investigational drug (allantoin, metronidazole, dexamethasone);
* Had used illicit drugs or had abused alcohol;
* Had a history of illness, or behavior (e.g., depression, psychosis) that in the opinion of the investigator might confound the results of the study or pose an additional risk in participating in the study;
* Women who were pregnant, and women who were of childbearing potential and not using method of birth control;
* Had participated in another clinical drug trial within the last 3 months;
* Were not agreed to participate the clinical trial by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Time to achieve recovery of both upper and lower GI function as measured by a composite endpoint of time to the first bowel movement and time to tolerate first solid food. This endpoint is referred to as GI2. | 7d

SECONDARY OUTCOMES:
Time to ready for discharge | 7 days
Time to the first flatus | 7 days
Comparison between the 2 groups of analgesics (morphine) dose | 7 days
peritoneal exudate volume of 72 hours after operation | 3 days
C reactive protein changes from baseline | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ying-jiang Ye, professor, Principal Investigator — Peking University People's Hospital
Locations (1):
- Center for Drug Clinical Research, Shanghai University of Chinese Medicine, Shanghai, Shanghai Municipality, China